CLINICAL TRIAL: NCT04813341
Title: Effectiveness of Mat Pilates and Aerobic Training on Fatigue Levels of Postpartum Females
Brief Title: Effectiveness of Mat Pilates and Aerobic Training on Fatigue and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/00844 Rida Fatima
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Post Partum Depression
Keywords: Depression; Fatigue; low intensity Aerobic training; Mat-Pilates
MeSH Terms: conditions — Depression, Postpartum; Depression; Fatigue | interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates training (Experimental): Bridging, roll up, one leg circle (both ways); single straight leg stretches; double leg stretches; side kick up and down; side kick circles
  Interventions: Other: Pilates training
- Aerobic Training (Active Comparator): WALKING: 10 mint brisk walk excluding warm up and cool down in 5 days/ week STATIONARY CYCLE: for 10 mints, 5 days/ week
  SITTING EERCISES:
  Chest stretch: ask to hold for 5 seconds and perform 5 repetitions Upper body twist: ask to cross the arms against chest and hold for 5 seconds, perform 5 repetitions Hip marching: Ask the client to sit on chair with arm rest and lift each of her leg 5 times
  BALANCE EXERCISES:
  Sideways walking: ask to perform 10 steps on each way (side to side), 5 days/week.
  Heel to Toe walk: perform at least 5 steps and increase gradually in each repetition, 5days/ week Step up and down: Ask to step up and down on given surface, 5 repetitions on each leg, 5 days/ week.
  Interventions: Other: Aerobic Training

INTERVENTIONS:
Other: Pilates training — Bridging, roll up, one leg circle (both ways); single straight leg stretches; double leg stretches; side kick up and down; side kick circles. The participant will be instructed to perform 3-5 repetitions of these movements at the start, and to add two more repetitions for each movement every week until the end of the intervention.
  Arms: Pilates training
Other: Aerobic Training — WALKING: 10 mint brisk walk excluding warm up and cool down in 5 days/ week STATIONARY CYCLE: for 10 mints, 5 days/ week
  SITTING EERCISES:
  Chest stretch: ask to hold for 5 seconds and perform 5 repetitions Upper body twist: ask to cross the arms against chest and hold for 5 seconds, perform 5 repetitions Hip marching: Ask the client to sit on chair with arm rest and lift each of her leg 5 times
  BALANCE EXERCISES:
  Sideways walking: ask to perform 10 steps on each way (side to side), 5 days/week.
  Heel to Toe walk: perform at least 5 steps and increase gradually in each repetition, 5days/ week Step up and down: Ask to step up and down on given surface, 5 repetitions on each leg, 5 days/ week.
  Arms: Aerobic Training

SUMMARY:
The aim is to see fatigue and depression levels in postpartum females and to evaluate ho two well-known exercises, Mat Pilates and Aerobic training can help to reduce the fatigue levels in postpartum females

DETAILED DESCRIPTION:
The aim is to see fatigue and depression levels in postpartum females and to evaluate ho two well-known exercises, Mat Pilates and Aerobic training can help to reduce the fatigue levels in postpartum females. In this study, the researcher will also compare the effects of Mat Pilates and Aerobic training on fatigue and depression levels among postpartum females.

ELIGIBILITY:
Inclusion Criteria:

* Vaginal delivery
* Singleton pregnancy

Exclusion Criteria:

* Caesarean delivery
* Vacuum-assisted delivery
* Sexually Transmitted Diseases
* Menopause females
* Any condition regarding Obstetrics & Gynecology
* Any physical or mental illness

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Multidimensional Fatigue Inventory | 6 weeks
  The MFI-20 is a self-report of 20-item scale designed to evaluate five dimensions of fatigue: general fatigue, physical fatigue, reduced motivation, reduced activity and mental fatigue. By limiting the length of questionnaire, developers hoped to accommodate those individuals who might find larger measures especially tiring in obtaining multiple facets of fatigue. The internal consistency of MFI-20 is ranging from .53 to .93.
Edinburgh Postnatal Depression Scale | 6 weeks
  EPDS developed for screening postpartum women in outpatient, home-visiting settings or at 6-8-week postpartum examination. It consists of 10 questions for postnatal period which reliably identifies women at risk of developing depression. The sensitivity and specificity of EPDS is 70-85%.

CONTACTS AND LOCATIONS:
Overall Officials: Anam Aftab, Phd*, Principal Investigator — Riphah college of rehabilitation and allied health sciences - Rawalpindi
Locations (1):
- Anmol Hospital Phalia, Jhelum, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No